CLINICAL TRIAL: NCT01802372
Title: Task Shifting and Blood Pressure Control in Ghana: A Cluster-Randomized Trial
Brief Title: Task Shifting and Blood Pressure Control in Ghana
Acronym: TASSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-01631; 1U01HL114198-01 (NIH)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Hypertension; High Blood Pressure; Cardiovascular Diseases
Keywords: Hypertension; High Blood Pressure; Cardiovascular Diseases; Health Insurance Coverage; Low income countries; Ghana; Low resource settings; Comparative Effectiveness; Global Health
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO CVD Risk Assessment package (Active Comparator): Arm#1 (Intervention Group): Provided Ghana's National Health Insurance and the WHO CVD Risk Assessment package for 12 months.
  Interventions: Behavioral: WHO CVD risk assessment package
- Health Insurance only (Sham Comparator): Arm#2 (Control group): Provided Ghana's National Health Insurance for 12 months, brief behavioral counseling at baseline,and usual care.
  Interventions: Behavioral: Health Insurance only

INTERVENTIONS:
Behavioral: WHO CVD risk assessment package — Arm#1 (Intervention Group): Provided Ghana's National Health insurance and the WHO CVD Risk Assessment package for 12 months.
  Arms: WHO CVD Risk Assessment package
Behavioral: Health Insurance only — Arm#2 (Control group): Provided Ghana's National Health Insurance for 12 months, brief behavioral counseling at baseline, and usual care.
  Arms: Health Insurance only

SUMMARY:
The goal of this study is to evaluate the comparative effectiveness of the World Health Organization Package targeted at Cardiovascular (CV) risk assessment and hypertension control, delivered by Community Health Nurses as part of Ghana's Community based Health Planning and Services program, versus provision of health insurance coverage, on blood pressure reduction. Findings from this study will provide policy makers and other stakeholders needed information to recommend efficient cost-effective policy with regards to comprehensive CV risk reduction in patients with hypertension in low resource settings.

DETAILED DESCRIPTION:
Countries in sub-Saharan Africa (SSA) are experiencing an epidemic of cardiovascular disease (CVD) propelled by rapidly increasing rates of hypertension. Barriers to hypertension control in SSA include poor access to care and high out-of-pocket costs. Although SSA bears 24% of the global disease burden, it has only 3% of the global health workforce. Given such limited resources, cost-effective strategies, such as task shifting, are needed to mitigate the rising CVD epidemic in SSA. Ghana, a country in SSA with an established community health worker program integrated within a national health insurance scheme provides an ideal platform to evaluate implementation of the World Health Organization (WHO) task-shifting strategy. This study will evaluate the comparative effectiveness of the implementation of the WHO Package targeted at CV risk assessment versus provision of health insurance coverage,on blood pressure (BP) reduction.

Using a cluster randomized design, 32 community health centers (CHCs) and district hospitals in Ghana will be randomized to either the intervention group (16 CHCs) or the control group (16 CHCs). A total of 640 patients with uncomplicated hypertension (BP 140-179/90-99 mm Hg and absence of target organ damage) will be enrolled in this study (20 patients per CHC). The intervention consists of WHO Package of CV risk assessment, patient education, initiation and titration of antihypertensive medications, behavioral counseling on lifestyle behaviors, and medication adherence every three months for 12 months. The primary outcome is the mean change in systolic BP from baseline to 12 months. The secondary outcomes are rates of BP control at 12 months; levels of physical activity, percent change in weight, and dietary intake of fruits and vegetables at 12 months; and sustainability of intervention effects at 24 months. All outcomes will be assessed at baseline, six months and 12 months. Trained community health nurses will deliver the intervention as part of Ghana's community-based health planning and services (CHPS) program. Findings from this study will provide policy makers and other stakeholders needed information to recommend scalable and cost-effective policy with respect to comprehensive CV risk reduction and hypertension control in resource-poor settings.

ELIGIBILITY:
Inclusion Criteria:

* Health facility Inclusion: Participating health facilities will be selected from areas that are geographically distant from one another with equal urban/rural mix in the Ashanti Region, which has 170 community health centers. Of these, we will recruit 32 for this study. Eligible facilities must have at least one community health nurse employed in the CHPS program; be a certified National Health Insurance Scheme (NHIS) provider; and have basic capability for blood tests.
* Patient Inclusion: To be eligible for the study, patients must fulfill the following criteria: a) are registered to receive care at the health center; b) are adults age 40 years and older; c) have BP 140-179/90-100 mm Hg and are not on treatment for hypertension; and c) can provide informed consent. Given low literacy levels, consent will be provided both verbally and in written form.

Exclusion Criteria:

-Patients will be excluded if they have: a) previous diagnosis of diabetes, coronary artery disease, transient ischemic attacks, stroke, heart failure, or angina: b) BP>180/100 mm Hg; c) positive urine dipstick for protein; d) are pregnant; and e) unable to comply with the follow-up requirements or provide informed consent. Patients with history of transient ischemic attacks (TIAs), stroke, heart failure, diabetes, angina, claudication, and BP>180/100 mm Hg will be referred to the district hospitals for further management.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Mean change in systolic Blood Pressure (BP) | Baseline to 12 months
  BP control is defined as BP<140/90

SECONDARY OUTCOMES:
Physical activity levels,change in weight,dietary intake of fruits and vegetables | 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gbenga Ogedegbe, MD, MS, MPH, Principal Investigator — NYU Langone Medical Center
Locations (1):
- Kwame Nkrumah University of Science and Technology, Kumasi, Ghana

REFERENCES:
- [Derived] Gyamfi J, Allegrante JP, Iwelunmor J, Williams O, Plange-Rhule J, Blackstone S, Ntim M, Apusiga K, Peprah E, Ogedegbe G. Application of the Consolidated Framework for Implementation Research to examine nurses' perception of the task shifting strategy for hypertension control trial in Ghana. BMC Health Serv Res. 2020 Jan 29;20(1):65. doi: 10.1186/s12913-020-4912-5. PMID 31996195
- [Derived] Ogedegbe G, Plange-Rhule J, Gyamfi J, Chaplin W, Ntim M, Apusiga K, Iwelunmor J, Awudzi KY, Quakyi KN, Mogaverro J, Khurshid K, Tayo B, Cooper R. Health insurance coverage with or without a nurse-led task shifting strategy for hypertension control: A pragmatic cluster randomized trial in Ghana. PLoS Med. 2018 May 1;15(5):e1002561. doi: 10.1371/journal.pmed.1002561. eCollection 2018 May. PMID 29715303
- [Derived] Gyamfi J, Plange-Rhule J, Iwelunmor J, Lee D, Blackstone SR, Mitchell A, Ntim M, Apusiga K, Tayo B, Yeboah-Awudzi K, Cooper R, Ogedegbe G. Training nurses in task-shifting strategies for the management and control of hypertension in Ghana: a mixed-methods study. BMC Health Serv Res. 2017 Feb 2;17(1):104. doi: 10.1186/s12913-017-2026-5. PMID 28148255
- [Derived] Ogedegbe G, Plange-Rhule J, Gyamfi J, Chaplin W, Ntim M, Apusiga K, Khurshid K, Cooper R. A cluster-randomized trial of task shifting and blood pressure control in Ghana: study protocol. Implement Sci. 2014 Jun 12;9:73. doi: 10.1186/1748-5908-9-73. PMID 24923300